CLINICAL TRIAL: NCT02676258
Title: A Prospective Randomized Controlled Study to Evaluate the Clinical Performance of Si-Hy Silicone Hydrogel Soft Contact Lens
Brief Title: Clinical Comparison of Two Daily Disposable Silicone Hydrogel Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visco Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1030313M
Record Dates: First submitted 2016-01-30; First posted 2016-02-08 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Myopia
Keywords: silicone hydrogel daily disposable soft contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Si-Hy soft contact lens (Experimental): olifilon B daily disposable soft contact lens
  Interventions: Device: Si-Hy (olifilcon B)
- Vistakon soft contact lens (Active Comparator): narafilcon A daily disposable soft contact lens
  Interventions: Device: Vistakon (narafilcon A)

INTERVENTIONS:
Device: Si-Hy (olifilcon B) — Wear Si-Hy silicone hydrgel soft contact lens for 3 months
  Arms: Si-Hy soft contact lens
Device: Vistakon (narafilcon A) — Wear Vistakon soft contact lens for 3 months
  Arms: Vistakon soft contact lens

SUMMARY:
The objective of this study is to evaluate a new daily disposable silicone hydrogel soft contact lens by comparing to an existing daily disposable soft contact lens.

DETAILED DESCRIPTION:
This study is designed to evaluate the performance of the olifilcon B contact lens to demonstrate substantial equivalence to the narafilcon A for regulatory requirement.

ELIGIBILITY:
Inclusion Criteria:

* Subject should have normal eyes and use no ocular medications
* Subject with -1.00 to -10.00 D myopia, less than 2.00 D astigmatism
* VA correctable to Log MAR 0.1 or better.
* Willing to comply with all study procedures and be available for the duration of the study.
* Provide signed and dated informed consent form.

Exclusion Criteria:

* Subjects have history of allergies that would contraindicate "normal" contact lens wear.
* Subjects have other active ocular or systemic disease such as, but not limited to : anterior uveitis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermas, keratoconus or type II diabetes.
* Subjects have medications that would contraindicate contact lens wear.
* Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the next 3 month.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any active participation in another clinical trial within 30 days prior to this study.
* The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates or fungal infections.
* A history of papillary conjunctivitis that has interfered with contact lens wear.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | over all follow-up visits for 3 month study period
  logMAR visual acuity (VA) over all visits.

SECONDARY OUTCOMES:
Any Slit Lamp Finding > Grade 2 | over all follow-up visits for the 3 month study period
  All dispensed eyes over all follow-up visits. Measured on a scale of 0-4 with 0=no findings and 4=sever findings.
Subjective Response to Comfort, symptoms and complaints | over all follow-up visits for the 3 month study period
  subjective ratings of comfort, symptom and complaints using a scale of 0=severe stinging/Burning to 10=No stinging/Burning for each eye; 0 represented the least favorable rating and a 100 represented the most favorable rating.

CONTACTS AND LOCATIONS:
Overall Officials: Huey Chuan Cheng, MD MS, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- MayKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No